CLINICAL TRIAL: NCT03496792
Title: The Venous Distension Reflex and Orthostatic Hypertension
Acronym: OH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jian Cui, Associate Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00007397
Record Dates: First submitted 2018-02-15; First posted 2018-04-12 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Blood Pressure
Keywords: venous distension reflex

STUDY DESIGN:
Intervention Model Description: The investigators will examine if individuals with elevated standing blood pressure have a heightened VDR. Two groups of subjects, "BP elevated with standing" group and "BP maintained with standing" group will be examined for this experiment. The tilt + external pressure and tilt + no external pressure, or the limb occlusion + negative pressure and limb occlusion + no negative pressure trials will be performed in random order using a Latin Square design. Because the nature of the interventions, neither the subjects nor the investigators can be blinded to the interventions
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will not know trial intervention prior to data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Tilt + external pressure (Experimental): Tilt + external pressure on legs performed in both "BP elevated with standing" and "BP maintained with standing" groups.
  Interventions: Other: Tilt + external pressure
- Tilt + no external pressure (Placebo Comparator): Tilt + no external pressure performed in both "BP elevated with standing" and "BP maintained with standing" groups.
  Interventions: Other: Tilt + no external pressure.
- Limb occlusion + negative pressure (Experimental): Limb occlusion + negative pressure performed in both "BP elevated with standing" and "BP maintained with standing" groups.
  Interventions: Other: Limb occlusion + negative pressure
- Limb occlusion + no negative pressure (Placebo Comparator): Limb occlusion + no negative pressure performed in both "BP elevated with standing" and "BP maintained with standing" groups.
  Interventions: Other: Limb occlusion + no negative pressure

INTERVENTIONS:
Other: Tilt + external pressure — In Visit 1, the anti-shock trousers will be inflated to 20, 40, or 60 mmHg. BP will be measured 3 times from the brachial artery. Then the table will be tilted head up to a maximum of 70o for up to 10 min, while BP will be measured from the brachial artery at 1 min intervals. The tilt table is returned to 0o and the resting supine baseline BP will be collected. Then, the anti-shock trousers will be inflated to a different pressure (20, 40, or 60 mmHg) and the head up tilt will be repeated. Repetitions at the various pressures will be performed in a random order with suitable resting intervals in between the tilting bouts.
  Arms: Tilt + external pressure
Other: Tilt + no external pressure. — In Visit 1, the anti-shock trousers will NOT be inflated. Auscultatory BP will be measured 3 times from the brachial artery. Thereafter, the table will be tilted head up to a maximum of 70o for up to 10 min, while BP will be measured from the brachial artery at 1 min intervals.
  Arms: Tilt + no external pressure
Other: Limb occlusion + negative pressure — In Visit 2, a cuff will be placed on the thigh of a leg that is sealed in an airtight pressure tank. After the cuff is inflated to 250 mmHg, the pressure in the tank will be reduced to -100mmHg for 2 minutes. The application of negative pressure creates a suction effect on the leg, and leads to an overall increase in pressure gradient across the blood vessel wall and induces vascular distension.
  Arms: Limb occlusion + negative pressure
Other: Limb occlusion + no negative pressure — In Visit 2, a cuff will be placed on the thigh of a leg that is sealed in an airtight pressure tank. The cuff is inflated to 250 mmHg for 2 minutes, but the pressure in the tank is not changed.
  Arms: Limb occlusion + no negative pressure

SUMMARY:
This research is being done to find out whether distension of veins in legs will cause a rise in blood pressure (orthostatic hypertension).

DETAILED DESCRIPTION:
In humans, two-thirds of the blood volume is contained within the venous vasculature. Because of this, changes in peripheral blood volume and alterations in the mechanical properties of peripheral veins can greatly impact cardiac filling, cardiac output and blood pressure (BP) responses to physiologic stress. Work from our laboratory over the past seven years has shown that local upper limb venous distension via volume infusion into an occluded arm (i.e. volume infusion model) or applying negative pressure to an occluded leg (limb suction experimental model) leads to an acute and dramatic increase in Muscle Sympathetic Nerve Activity (MSNA; an index of sympathetic activity directed to skeletal muscle) and BP in humans. Since this venous distension reflex (VDR) differs physiologically from the other reflex systems, and since this system may play a critical role in orthostatic BP control, we believe that it is a significant area of study.

The investigators speculate that VDR from lower limbs contributes to the autonomic adjustment to orthostatic stress. To examine the VDR in lower limbs, an arterial occlusion cuff on the mid-thigh was inflated (250 mm mercury; Hg). Then, limb suction (-100 mmHg) was applied ~10-15 cm below the level of arterial occlusion (i.e. below the knee). MSNA was measured in the opposite control limb. When suction was applied below the level of arterial occlusion (i.e. occlusion + suction), both MSNA and mean arterial BP (MAP) increased. In control trials, arterial occlusion without limb suction (i.e. occlusion alone) did not increase MSNA. Plethysmographic data showed calf circumference increased without detectable arterial pulsations. Pilot data suggest that the fluid shifts from the occluded but non-depressurized zone of the limb (i.e. between the cuff and knee) into the occluded and depressurized region of the limb within the tank. Thus, the results suggest that the VDR was engaged with this limb suction experimental model.

These experimental models "selectively" alter peripheral venous volume as the investigators measure sympathetic reflex responses. This approach is innovative and allows examination of a previously overlooked autonomic reflex in conscious humans. If these studies confirm the hypotheses, the obtained data would challenge the present teaching regarding how the sympathetic nervous system is engaged in humans during postural stress.

In ~2.5-10% of the population, BP rises as the person stands. This has been termed orthostatic hypertension, and is different from the "normal" sustained BP response when a person stands. The incidence of orthostatic hypertension may increase with aging (~2.4% for 45-64 years old and ~8.7% for >70 years old). Orthostatic hypertension is a risk factor for the development of stroke, left ventricular hypertrophy, and chronic kidney disease. It is unclear why BP rises with standing in some individuals. Some investigators have speculated that orthostatic hypertension is due to exaggerated baroreceptor withdrawal with standing. Others have speculated that this response is due to an increase in sympathetic output. It has been noted that some patients with orthostatic hypertension have increased venous pooling in their lower legs. Based these data, the investigators postulate that heightened engagement of the VDR reflexly increases MSNA and also serves to reset the aortic baroreflex. In this protocol, the investigators will determine if the MSNA response to leg suction is heightened in the individuals with elevated standing BP, and examine if the baroreflex is altered in these individuals. The investigators will also examine if external pressure on lower limbs, which limits the venous pooling in the lower limbs, will attenuate the increase in BP during standing in those individuals.

ELIGIBILITY:
Inclusion Criteria:

* Are capable of giving informed consent
* Are of any race or ethnicity
* Are fluent in written and spoken English
* Whose history and physical exam did not uncover any exclusion criteria
* Are 18 years of age

For subjects with elevated standing BP

* Systolic BP (SBP) during standing is at least 10 mmHg > the supine SBP
* Patients with a diagnosis of stage I hypertension without other chronic diseases may be INCLUDED

For normal subjects without elevated standing BP

* The change in SBP by standing is within ± 5 mmHg from the supine SBP
* Matched gender, similar age and BMI (within 10%) to participants with elevated standing BP
* Free of acute or chronic medical conditions

Exclusion Criteria:

* Age < 18 years of age
* Are a pregnant or nursing woman
* Are a prisoner or institutionalized individual or unable to consent
* Have chronic diseases (e.g. heart, lung, neuromuscular disease, or cancer) other than stage I hypertension
* Have orthostatic hypotension or a history of syncope
* Current smoker
* History of blood clots

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Muscle Sympathetic Nerve Activity (MSNA) in bursts/min or arbitrary units/min | Recorded continuously during Visit 2, the 4-5 hr Negative Pressure study visit.
  MSNA provides direct recordings of sympathetic nerve activity directed to blood vessels in skeletal muscle.

SECONDARY OUTCOMES:
Blood pressure in mmHg | Recorded continuously during the 4-5 hr visit.
  Cuffs placed on a finger and arm will monitor blood pressure.
Heart rate in beats per minute | Recorded continuously during the 4-5 hr visit.
  Electrocardiogram (ECG) patches attached to a Cardiocap will monitor heart rate.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Cui, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Cui J, Blaha C, Herr MD, Drew RC, Muller MD, Sinoway LI. Limb suction evoked during arterial occlusion causes systemic sympathetic activity in humans. Am J Physiol Regul Integr Comp Physiol. 2015 Sep;309(5):R482-8. doi: 10.1152/ajpregu.00117.2015. Epub 2015 Jul 1. PMID 26136530
- [Background] Cui J, Gao Z, Blaha C, Herr MD, Mast J, Sinoway LI. Distension of central great vein decreases sympathetic outflow in humans. Am J Physiol Heart Circ Physiol. 2013 Aug 1;305(3):H378-85. doi: 10.1152/ajpheart.00019.2013. Epub 2013 May 31. PMID 23729210
- [Background] Cui J, Leuenberger UA, Gao Z, Sinoway LI. Sympathetic and cardiovascular responses to venous distension in an occluded limb. Am J Physiol Regul Integr Comp Physiol. 2011 Dec;301(6):R1831-7. doi: 10.1152/ajpregu.00170.2011. Epub 2011 Sep 21. PMID 21940404
- [Background] Cui J, McQuillan PM, Blaha C, Kunselman AR, Sinoway LI. Limb venous distension evokes sympathetic activation via stimulation of the limb afferents in humans. Am J Physiol Heart Circ Physiol. 2012 Aug 15;303(4):H457-63. doi: 10.1152/ajpheart.00236.2012. Epub 2012 Jun 15. PMID 22707559
- [Background] Cui J, McQuillan P, Moradkhan R, Pagana C, Sinoway LI. Sympathetic responses during saline infusion into the veins of an occluded limb. J Physiol. 2009 Jul 15;587(Pt 14):3619-28. doi: 10.1113/jphysiol.2009.173237. Epub 2009 May 26. PMID 19470776
- [Background] Kario K. Orthostatic hypertension-a new haemodynamic cardiovascular risk factor. Nat Rev Nephrol. 2013 Dec;9(12):726-38. doi: 10.1038/nrneph.2013.224. Epub 2013 Nov 5. PMID 24189649